CLINICAL TRIAL: NCT00572611
Title: A Phase I Study to Investigate the Absorption, Metabolism and Excretion of [14C]-Bilastine Following Oral Administration to Healthy Volunteers
Brief Title: Human Mass Balance Study With Bilastine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: Charles River Clinical Services Edinburgh Ltd and CR Laboratories Preclinical Services Ltd (Unknown); MDS Pharma Services Switzerland AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BILA 459-13; EudraCT Number: 2007-003373-12; CR Study Number: 186781
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Mass Balance; Metabolism; Absorption; Excretion; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Single oral dose of 20 mg [14C]-bilastine
  Interventions: Drug: [14C]-bilastine

INTERVENTIONS:
Drug: [14C]-bilastine — Single oral dose of 20 mg [14C]-bilastine. 1 capsule. 1 day dosing only

SUMMARY:
The primary objective of the study is to define the absorption and excretion kinetics of bilastine in man following oral administration, and to investigate the nature of the metabolites present in plasma and excreta. The secondary objective of the study is to assess the safety and tolerability of bilastine

DETAILED DESCRIPTION:
Primary Endpoints are: Whole blood and plasma concentrations of total radioactivity and parent drug. Urine and faecal recovery of total radioactivity. Characterisation and identification of metabolites in plasma, urine and faeces.

ELIGIBILITY:
Inclusion Criteria:

* No clinically important abnormal physical findings.
* No clinically significant abnormalities in the results of laboratory evaluation.
* Normal ECG.
* Normal supine blood pressure and heart rate.
* Body weight between 50 and 100 kg and body mass index between 18 and 30 kg/m2.
* Able to communicate well with the investigator and to comply with the requirements of the entire study.
* Provision of written informed consent to participate.
* Subjects must agree to use an adequate method of contraception during the study and for 12 weeks after dosing.
* Subjects must have a negative urine screen for drugs of abuse.
* Subjects must have a regular bowel habit.

Exclusion Criteria:

* Administration of any IMP within 12 weeks before entry to the study.
* Use of any prescribed medication or St John's Wort within 14 days or OTC medication within 5 days of dosing.
* Existence of any surgical or medical condition which, in the judgement of the investigator, might interfere with the absorption, distribution, metabolism or excretion of the IMP.
* History of any drug or alcohol abuse in the past 2 years, or alcohol consumption greater than 21 units per week.
* Presence or history of allergy requiring treatment.
* Hayfever is allowed unless it is active or has required treatment within the previous 2 months.
* Donation or loss of greater than 400 mL of blood within 12 weeks before entry to the study.
* Serious adverse reaction or serious hypersensitivity to any drug.
* Presence of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab) or HIV 1 or HIV 2 antibodies at screening.
* Administration of radiolabelled substances or exposure to significant radiation (eg serial x-ray or CT scans, barium meal etc) within the past 12 months.
* Any ECG abnormality at screening (including QTc intervals of >430 ms).
* Past medical history of clinically significant ECG abnormalities, or a family history of a prolonged QT interval syndrome.
* Abnormal diet or substantial changes in eating habits within 30 days prior to study initiation.
* Treatment with any known enzyme altering agents (barbiturates, phenothiazines, cimetidine, etc.) within 2 months prior to or during the study.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Whole blood and plasma concentrations of total radioactivity and parent drug | 168-216 h after dosing, depending on the radioactivity recovery
Urine and faecal recovery of total radioactivity | 168-216 h after dosing, depending on the radioactivity recovery
Characterisation and identification of metabolites in plasma, urine and faeces | 168-216 h after dosing, depending on the radioactivity recovery

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Mair, MD, Principal Investigator — Syneos Health; Lindsay McGregor, Study Director — Syneos Health
Locations (1):
- Charles River Laboratories Clinical Services Ltd, Origo Centre, Riccarton, Edinburgh, United Kingdom

REFERENCES:
- [Background] Lucero ML, Gonzalo A, Mumford R, Betanzos M, Alejandro A. An overview of bilastine metabolism during preclinical investigations. Drug Chem Toxicol. 2012 Jun;35 Suppl 1:18-24. doi: 10.3109/01480545.2012.682651. PMID 22616812
- [Background] Lucero ML, Patterson AB. Whole-body tissue distribution of total radioactivity in rats after oral administration of [(1)(4)C]-bilastine. Drug Chem Toxicol. 2012 Jun;35 Suppl 1:1-7. doi: 10.3109/01480545.2012.682650. PMID 22616810